CLINICAL TRIAL: NCT05920096
Title: Feasibility Assessment of a Diabetes Specialist Nurse-led Multi-component Smoking Cessation Intervention for Individuals Living With Diabetes
Brief Title: Feasibility of a Diabetes Specialist Nurse-led Smoking Cessation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Joseph Grech, Principal Investigator, University of Malta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V_15062020 8618
Record Dates: First submitted 2023-05-31; First posted 2023-06-27 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus; Tobacco Use Cessation
Keywords: Intervention Study; Feasibility Studies; Acceptability; Information Motivation Behavioral Skills Model; Counselling; Smoking Cessation Agents; 5A's Framework
MeSH Terms: conditions — Diabetes Mellitus; Tobacco Use Cessation | interventions — Health Promotion; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A diabetes specialist nurse-led multi-component smoking cessation intervention tailored for individuals with diabetes based on evidence and theory and guided by the 5A's and 5R's framework for smoking cessation The intervention consists of three to four (30-60 minutes) smoking cessation support sessions which are to be delivered by the two diabetes specialist nurses at the Diabetes Education Unit during the study period (12 weeks). As part of the first session, participants will also be shown three very brief video clips in which a person living with diabetes explains the serious health problems he suffered from (when smoking and having diabetes). Participants will also receive a six-week supply of Nicotine Replacement Therapy (NRT) - nicotine patch and/or nicotine spray.
  Interventions: Other: Diabetes specialist nurse-led multi-component smoking cessation intervention
- Control (Active Comparator): Active referral to the Health Promotion and Disease Prevention Directorate's one-to-one general stop-smoking service. This counseling service is provided every fortnight within Mosta, Floriana, or Paola health centres. The number of counseling sessions (lasting around 20 minutes each) provided during the study period (12 weeks) will be based on the client's needs.
  Interventions: Behavioral: Health Promotion and Disease Prevention Directorate's one-to-one smoking cessation service (standard care)

INTERVENTIONS:
Other: Diabetes specialist nurse-led multi-component smoking cessation intervention — Aims to:
  * inform participants on the association between smoking and diabetic complications;
  * motivate and encourage smokers to quit;
  * support participants in using the appropriate behavioural skills to quit smoking and avoid relapse.
  In the first session, the participants will be supported to set a Target Quit Date (TQD) within two weeks. Participants will be followed up within a week (or two weeks max.) from their TQD. Those who report having not smoked (for ≥24 hours from the time of assessment) will be provided with a final follow-up session within five weeks from their set TQD (three sessions in total). Conversely, those who report still smoking will be encouraged to set another TQD and will be seen again in one (or two weeks max.) and five weeks from their new TQD (four sessions in total). The participants will also receive a six-week supply of Nicotine Replacement Therapy (NRT) nicotine patch and/or spray to use for a few days prior to their TQD and on quitting.
  Arms: Intervention
Behavioral: Health Promotion and Disease Prevention Directorate's one-to-one smoking cessation service (standard care) — A behavioral smoking cessation intervention based on motivational interviewing and delivered by trained tobacco cessation facilitators within community health centres. Participants will be provided with 20-minute counseling sessions based on their needs.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to assess the feasibility and acceptability of a multi-component smoking cessation intervention for individuals living with diabetes which is delivered by diabetes specialist nurses. The main question it aims to answer is:

Is a diabetes specialist nurse-led multi-component smoking cessation intervention tailored for persons living with diabetes who smoke feasible and acceptable among the providers and the participants, the individuals with diabetes?

Eligible individuals living with diabetes who smoke will be asked to participate in a feasibility study lasting twelve weeks. The participants will be allocated at random either to the diabetes specialist nurse-led multi-component smoking cessation intervention, or to standard care - an active referral to the Health Promotion and Disease Prevention Directorate's one-to-one smoking cessation service. The multi-component smoking cessation intervention will be provided by the diabetes specialist nurses at the Diabetes Education Unit at Mater Dei Hospital. The Health Promotion and Disease Prevention Directorate's one-to-one smoking cessation service is provided by tobacco cessation facilitators within the health centres of Mosta, Floriana, and Paola. Both interventions will help participants re-consider their smoking habits and support them to quit smoking, free of charge.

Primarily the researchers will:

* assess the feasibility of a largescale randomized controlled trial, by analyzing the recruitment and study uptake, and the nurses' perceived challenges and facilitators to implementation;
* and assess the acceptability of the intervention, by analyzing the nurses' feedback and the participants' satisfaction with and perceived usefulness of the smoking cessation intervention provided, in comparison to the satisfaction with standard care - the Health Promotion and Disease Prevention Directorate's one-to-one smoking cessation service.

DETAILED DESCRIPTION:
BACKGROUND

Smoking cessation is an important aspect of diabetes management. Smoking worsens the cardiometabolic parameters of both individuals with type 1 and type 2 diabetes, significantly increasing the risk of various macro- and micro-vascular complications, and even death. Smoking cessation is associated with improved cardiometabolic values and a reduced risk of cardiovascular complications. However, evidence suggests that people living with diabetes may less likely quit smoking when compared to those without diabetes.

While the need for providing tailored smoking cessation support for those who have diabetes has been emphasized, evidence-based smoking cessation recommendations for such individuals are lacking. In addition, the literature suggests that diabetes educators tend to focus on other aspects of diabetes management, rather than tobacco use. Diabetes educators have reported feeling inadequately prepared in discussing smoking cessation amongst individuals with diabetes lacking motivation and time to do so.

STUDY AIM AND OBJECTIVES

The aim of this randomized controlled feasibility study is to establish the feasibility and acceptability of a diabetes specialist nurse-led smoking cessation intervention, based on evidence and theory, tailored for people living with diabetes.

The primary objectives are to:

* assess the feasibility of a large-scale randomized controlled trial, by analyzing the recruitment and study uptake, and the nurses' perceived challenges and facilitators to implementation;
* and assess the acceptability of the intervention, by analyzing the participants' satisfaction with and perceived usefulness of the smoking cessation support provided, and the nurses' feedback.

The secondary objectives are to:

* compare the participants' satisfaction with and perceived usefulness of the smoking cessation support provided to standard care - the provision of general smoking cessation support;
* undergo a preliminary process evaluation, by assessing whether the intervention was delivered as intended and exploring the intervention's functioning;
* and determine the preliminary evidence of the intervention's effectiveness, by comparing the smoking cessation rates achieved in the intervention group to the control group (standard care).

METHODS

Design

An open-label, two-arm randomized controlled trial.

Participants

Participants (individuals with diabetes) will be recruited from the Diabetes Education Unit and the Diabetes and Endocrine Centre (MOP2) at Mater Dei Hospital in Malta. The diabetes specialist nurses at the Diabetes Education Unit and the diabetologists and health care professionals at MOP2 will be identifying attending smokers, recruiting those who are interested to the study. Posters and flyers will also be present at MOP2 so that participants can also self-refer to the study. For feasibility studies, 30 to 60 participants per group have been suggested. Given that the sample size decision must also take into consideration the resources required and the time available, this study aims to recruit between 80 to 100 participants in total over a 12 month-period.

Implementation and data collection methods

The Principal Investigator (PI) will screen all recruited patients to determine eligibility and obtain informed consent. Demographic data, the participants' perceived health status, their diabetes and smoking profiles, and reported feelings in the past week will be assessed using a questionnaire. Exhaled carbon monoxide will also be measured using the Bedfont piCO™ Smokerlyzer®. Participants will then be randomly allocated to the intervention or control arm on a 1:1 ratio using a computer-generated random block length, which will be concealed to the PI.

The participants assigned to the intervention group will receive a tailored smoking cessation intervention for individuals with diabetes based on evidence and theory and guided by the 5A's (Ask, Advise, Assess, Assist and Arrange) and 5R's (Relevance, Risks, Rewards, Roadblocks, and Repetition) framework for smoking cessation. This will consist of three to four (30-60 minutes) smoking cessation support sessions which will be provided by the two diabetes specialist nurses at the Diabetes Education Unit during the study period (12 weeks). As part of the first session, participants will also be shown three very brief video clips in which a person living with diabetes explains the serious health problems he suffered from (when smoking and having diabetes). Participants will also receive a six-week supply of Nicotine Replacement Therapy (NRT) - nicotine patch and/or nicotine spray. Conversely, the participants who are assigned to the control group will be actively referred to the Health Promotion and Disease Prevention Directorate's one-to-one smoking cessation service which is provided by tobacco cessation facilitators at Mosta, Floriana, or Paola health centres. These participants will be provided with a number of smoking cessation sessions (20 minutes each) based on their needs, provided every fortnight during the 12-week study period.

To help capture fidelity, all the sessions provided by the diabetes specialist nurses will be audio-recorded with consent. The nurses, who will provide the experimental intervention, will also be asked to document the following information per participant:

* the number (and duration) of the sessions provided (and the total time period [in weeks] during which the sessions were provided);
* whether the participant opted not to see the informational video clips (with reasons);
* whether the participant agreed to attempt to quit smoking (by setting a Target Quit Date, TQD) at their first session, (and subsequent session if still smoking), with reasons for not wanting to;
* provision of the 5R's intervention at the first session;
* non-attendance (and reasons);
* the amount of NRT provided (and returned);
* reported use of NRT (with reasons if a participant reports not using it) - including the total number of days of the nicotine patch and/or spray use (and the average use of the nicotine spray/day) during the first week following the TQD (and the subsequent TQD for those who agree to reattempt quitting), and in the next four weeks;
* any problems encountered (such as side effects on using NRT, identified mental health issues, issues with managing diabetes, and any referrals, [including reasons for refusing support]).

The tobacco cessation officer at the Health Promotion and Disease Prevention Directorate will also be asked to take note of the number of sessions provided (including the total time period during which the sessions were provided) and any dropouts (with reasons).

At the end of the study period, all participants will be asked to fill in the end-of-study questionnaire (to assess smoking and measure abstinence, characterize the support utilized, and investigate the participants' satisfaction with and perceived usefulness of the smoking cessation intervention provided). For those who report quitting smoking (for at least seven days prior to assessment), biochemical verification of tobacco abstinence will be carried out by using the Bedfont piCO™ Smokerlyzer®, and analyzing a urine sample for cotinine exposure using a multilevel lateral flow immunoassays urine test strip with a nominal 200 ng/mL cutoff.

Semi-structured interviews will also be carried out with a sample (15-20) of the study intervention participants to obtain feedback on the study intervention and to explore their quit attempts. Semi-structured interviews will also be carried out with the two diabetes specialist nurses to obtain feedback on the study intervention and to explore the facilitators and challenges to implementation.

Data analysis

Recruitment - The average number of participants recruited per month and the total time period taken to recruit all participants will be calculated. Reasons for ineligibility or for not consenting to participate to the study will be noted. The number of eligible individuals who accept to participate in the study out of those who show interest will be calculated with 95% Confidence Intervals (CIs).

Study questionnaires - Quantitative data, collected at baseline and at the end of the study period, will be analyzed per study group using descriptive statistics. For categorical data, frequencies and proportions/percentages will be used. Continuous data will be summarised using mean and standard deviation, or median and range or interquartile range. Qualitative data will be summarised by following the Applied Thematic Analysis (ATA) approach. The questionnaires' response rate at 12 weeks follow-up, the participants' satisfaction with and perceived usefulness of the smoking cessation intervention provided, and the smoking cessation outcomes, will also be reported using 95% CIs. Intention-to-treat analysis will be used; smokers who can not be reached or are lost to follow-up will be considered non-quitters and non-reducers. The baseline characteristics of those followed up and those lost to follow-up will be compared descriptively.

Interviews - The audio-recorded interviews will be transcribed verbatim, anonymized, and analyzed using ATA.

To provide a further understanding of the acceptability of the study intervention and its functioning as experienced by the study participants (individuals with diabetes) the quantitative and qualitative data will be compared for confirming, disconfirming, or expanding each other.

Audio recording of the provision of the study intervention - To assess fidelity, a random sample (20%) from all the audio recordings of the sessions provided by each provider will be selected. By using a checklist that outlines the study algorithm's components, the occurrence or non-occurrence of these steps will be scored for calculating the level of adherence. Any deviations from the study protocol will also be taken note of.

Intervention log - The rate of compliance to the provided interventions, i.e. the attendance rate to the scheduled sessions, and the reported use of NRT (intervention group only) will be noted. The latter includes the average percentage of days the nicotine patch and/or spray were used (and the average use of the nicotine spray/day) during the first week following the TQD (and the subsequent TQD for those who agree to reattempt quitting), and in the next four weeks. Reasons for non-attendance/not using NRT will be noted. The number of participants who opt not to see the informational video clips and the number of participants who do not want to set a TQD at their first session (and the subsequent session if they report still smoking) will also be noted (with reasons). In terms of resources utilized, the proportion of participants from the intervention group who are provided with the 5R's intervention, the total and average number of sessions provided (in both groups) and the average time period over which these are provided will be calculated. The average time taken to deliver the sessions in the intervention group will also be calculated. In addition, the total and average amount of NRT which are provided (taking note of any returned items) will be calculated (intervention group). Proportions/rates and means with standard deviation will be reported using 95% CIs. Any problems (including reported adverse events) identified by the nurses (and referrals) will be quantified. Participants who refuse additional support will be noted (with reasons).

Ethical clearance for this study was sought from the Faculty of Health Sciences Research Ethics Committee on behalf of the University Research Ethics Committee (UREC FORM V_15062020 8618)

ELIGIBILITY:
Inclusion Criteria:

* Living with type 1 or type 2 diabetes and attending the Diabetes Education Unit or the Diabetes and Endocrine Centre (MOP2) at Mater Dei Hospital on an outpatient basis
* Having smoked ≥100 cigarettes during his/her entire life and currently smoking (having at least smoked one tobacco product over the past 7 days)
* Being ≥ 18 years old
* Speaking and understanding English or Maltese
* Able to provide written informed consent

Exclusion Criteria:

* Not being able to provide informed consent (due to dementia, a learning disability, or a psychological disorder)
* Being pregnant or breastfeeding
* Unable to independently attend to the Diabetes Education Unit and the Mosta, Floriana, or Paola health centres in Malta during the 12-week study period
* Currently enrolled in another smoking cessation study/program or multi-behavioral program which also focuses on smoking cessation
* Enrolment of the investigator or the research collaborators, and their family members

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Feasibility (recruitment parameters) - recruitment rate | Baseline
  The average number of eligible participants recruited per month.
Feasibility (recruitment parameters) - the proportion of eligible smokers who indicate an interest in participating in the study from each source of recruitment | Baseline
  Sources of recruitment include: the diabetes education unit and the diabetes and endocrine centre [(MOP2) and self-referral (from posters and flyers present at the diabetes out-patients department).
Feasibility (recruitment parameters) - consent rate | Baseline
  The proportion of participants who consent to participate to the study out of the number of individuals who initially indicated an interest in participating and meet the eligibility criteria, including reasons for not consenting.
Feasibility (recruitment parameters) - the total time period of recruitment | Baseline
  Total time period (in months).
Feasibility (participation compliance) - participation rate in both groups | 12 weeks
  The proportion of participants who attend the scheduled sessions per group, with reasons for dropping out.
Feasibility (participation compliance) - the proportion/number of participants from the intervention group who opt not to see the informational video clips | 12 weeks
  The proportion/number of participants from the intervention group who opt not to see the informational video clips at their first session, with reasons.
Feasibility (participation compliance) - the proportion/number of participants from the intervention group who opt not to set a Target Quit Date (TQD) | 12 weeks
  The proportion/number of participants from the intervention group who opt not to set a TQD at their first session, with reasons.
Feasibility (participation compliance) - the proportion/number of continuing smokers from the intervention group who opt not to set a subsequent TQD | 12 weeks
  The proportion/number of continuing smokers from the intervention group who opt not to set a subsequent TQD at their second session, with reasons.
Feasibility (participation compliance) - reported use of Nicotine Replacement Therapy (NRT) on the TQD in the intervention group | 12 weeks
  The proportion of participants who report having used the nicotine patch and/or spray on their TQD (and on the subsequent TQD for continuing smokers), with reasons for not using it.
Feasibility (participation compliance) - average percentage of days of NRT use during the first week following the TQD in the intervention group | 12 weeks
  The average percentage of days the nicotine patch and/or spray were used during the first week following the TQD (and the subsequent set TQD among continuing smokers).
Feasibility (participation compliance) - average use of the nicotine spray per day during the first week following the TQD in the intervention group | 12 weeks
  The average number of times the nicotine spray was used per day during the first week following the TQD (and the subsequent TQD for continuing smokers).
Feasibility (participation compliance) - reported use of NRT during the final follow-up period in the intervention group | 12 weeks
  The proportion of participants who report having used the nicotine patch and/or spray during their final follow-up period, with reasons for not using it.
Feasibility (participation compliance) - average percentage of days of NRT use during the final follow-up period in the intervention group | 12 weeks
  The average percentage of days the nicotine patch and/or spray were used during the subsequent four weeks following one week from the TQD.
Feasibility (participation compliance) - average use of the nicotine spray per day during the final follow-up period in the intervention group | 12 weeks
  The average number of times the nicotine spray was used per day during the subsequent four weeks following one week from the TQD.
Feasibility (resources utilized) - average number of sessions provided in both groups | 12 weeks
  The average number of sessions provided per participant per group.
Feasibility (resources utilized) - average time period taken to provide smoking cessation support in both groups | 12 weeks
  The average time period (in weeks) per participant per group during which smoking cessation support was provided.
Feasibility (resources utilized) - average time taken to deliver the sessions in the intervention group | 12 weeks
  The average time (in minutes) taken to deliver the intervention sessions.
Feasibility (resources utilized) - provision of the 5R's intervention in the intervention group | 12 weeks
  The proportion/number of participants from the intervention group who were provided with the 5R's intervention.
Feasibility (resources utilized) - provision of NRT in the intervention group | 12 weeks
  The average amount of NRT provided per participant (taking note of any returned items).
Feasibility - response rate at 12 weeks follow-up | 12 weeks
  The proportion of participants who attend their 12-week post-intervention evaluation session (in the intervention and control groups). Participants who drop out from the study or are lost to follow-up at 12 weeks will be noted (with reasons).
Feasibility - number of problems (including reported adverse events when using NRT) identified by the nurses (intervention providers) and number of referrals to additional support services (e.g. psychotherapist, diabetologist). | through study completion, estimated at 12 months
  As logged by the nurses in carrying out the intervention. Participants who refuse additional support will be noted (with reasons).
Feasibility - nurses' (intervention providers) perceived challenges and facilitators to implementation (intervention group) | through study completion, estimated at 12 months
  As identified when conducting interviews with the nurses.
Acceptability - intervention group participants' satisfaction with the intervention provided (quantitative assessment) | 12 weeks
  By analyzing the results from the self-developed satisfaction questionnaire.
Acceptability - intervention group participants' satisfaction with the intervention provided (qualitative assessment) | 12 weeks
  As identified when conducting interviews with the participants.
Acceptability - intervention group participants' perceived usefulness of the intervention provided (quantitative assessment) | 12 weeks
  By analyzing the results from the self-developed perceived usefulness questionnaire.
Acceptability - intervention group participants' perceived usefulness of the intervention provided (qualitative assessment) | 12 weeks
  As identified when conducting interviews with the participants.
Acceptability - nurses' (intervention providers) satisfaction with the intervention | through study completion, estimated at 12 months
  As identified when conducting interviews with the nurses.

SECONDARY OUTCOMES:
Group comparison of the satisfaction with the intervention provided | 12 weeks
  Group comparison of the participants' satisfaction with the smoking cessation support provided as measured by the self-developed satisfaction questionnaire.
Group comparison of the perceived usefulness of the intervention provided | 12 weeks
  Group comparison of the results obtained from the self-developed questionnaire on the perceived usefulness of the smoking cessation intervention provided.
Preliminary process evaluation - intervention fidelity (intervention group) | through study completion, estimated at 12 months
  A random sample (20%) from all the audio recordings of the sessions provided by each provider will be selected. By using a checklist that outlines the study algorithm's components, the occurrence or non-occurrence of these steps will be scored for calculating the level of adherence. Any deviations from the study protocol will also be taken note of.
Preliminary process evaluation - exploring the intervention's functioning (intervention group) | 12 weeks
  As identified when conducting interviews with the participants.
Preliminary evidence of effectiveness - quit episode | 12 weeks
  Proportion of participants reporting a quit episode (intentionally have spent ≥24 hours not smoking or using smokeless/alternative products, e.g. electronic cigarettes) during the study period.
Preliminary evidence of effectiveness - floating abstinence | 12 weeks
  A reported 7-day point prevalence abstinence (from combustible tobacco products, smokeless tobacco products, and alternative products) at any time during the study period.
Preliminary evidence of effectiveness - change in average number of cigarettes smoked per day | 12 weeks
  The change in the average number of cigarettes smoked per day (amongst continuing smokers) per group at follow-up.
Preliminary evidence of effectiveness - point prevalence smoking abstinence at follow-up | 12 weeks
  The 7-day point prevalence abstinence (from combustible tobacco products, smokeless tobacco products, and alternative products) at follow-up, validated by measuring exhaled Carbon Monoxide (eCO) and additionally confirmed by using a multilevel lateral flow immunoassays urine test strip with a nominal 200 ng/mL cutoff for cotinine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Grech, PhD student, Principal Investigator — University of Malta
Locations (1):
- Diabetes Education Unit, Mater Dei Hospital, Msida, Malta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grech J, Norman IJ, Sammut R. Helping smokers with diabetes quit: A scoping review of the interventions utilised, and the challenges and barriers to smoking cessation. Prim Care Diabetes. 2023 Apr;17(2):119-128. doi: 10.1016/j.pcd.2023.01.005. Epub 2023 Jan 19. PMID 36681570
- [Background] Grech J, Norman IJ, Sammut R. Effectiveness of intensive stand-alone smoking cessation interventions for individuals with diabetes: A systematic review and intervention component analysis. Tob Induc Dis. 2023 May 10;21:57. doi: 10.18332/tid/162329. eCollection 2023. PMID 37181460
- [Background] Grech J, Norman IJ, Sammut R. Exploring the smoking cessation needs of individuals with diabetes using the Information-Motivation-Behavior Skills model. Tob Prev Cessat. 2024 Feb 2;10. doi: 10.18332/tpc/181366. eCollection 2024. PMID 38313659
- [Background] Grech J, Norman I, Azzopardi C, Grixti M, Sammut R. Assessing the feasibility and acceptability of a diabetes-specific nurse-led multicomponent smoking cessation intervention in diabetes education: study protocol for an open-label pragmatic randomised controlled trial. BMJ Open. 2024 Jun 19;14(6):e083235. doi: 10.1136/bmjopen-2023-083235. PMID 38904126
- [Background] Grech J, Norman IJ, Sammut R. Acceptability measures for evaluating smoking cessation interventions among individuals with diabetes. Public Health Pract (Oxf). 2024 Mar 2;7:100487. doi: 10.1016/j.puhip.2024.100487. eCollection 2024 Jun. PMID 38486708